CLINICAL TRIAL: NCT04920019
Title: Opioid Sparing Effect of Thoracic Epidural Analgesia for Open Upper Abdominal Surgery: Prospective Randomized Controlled Trial
Brief Title: Opioid Sparing Effect of Thoracic Epidural Analgesia for Open Upper Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Suwimon Tangwiwat, associate professor, Department of Anesthesiology, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: si 800/2020
Record Dates: First submitted 2021-05-21; First posted 2021-06-09 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Hepatoma; Pancreas Cancer
Keywords: open upper abdominal surgery; continuous epidural analgesia
MeSH Terms: conditions — Carcinoma, Hepatocellular; Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Group A: continuous epidural analgesia, Group B: no continuous epidural analsesia
Masking Description: Randomized group of patient is identified and sealed in envelope. Postoperative outcomes are assessed by Acute Pain Service nurse or resident.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic continuous epidural analgesia (Experimental): Thoracic continuous epidural analgesia at T7-8 or T8-9 combined with IV PCA fentanyl (bolus mode only 15 ug/bolus, 5 minutes lockout, 4 hours limit 200 ug).
  Multimodal analgesia Intraoperative : thoracic epidural infusion with 0.0625% bupivacaine with morphine 0.02 ug/ml 5 ml/h, morphine 2 mg epidurally are given.
  Postoperative: 0.0625% bupivacaine with morphine 0.02 ug/ml 5 ml/h is given combined with IV patient-controlled analgesia; bolus mode only, fentanyl 15 ug/bolus, lockout interval 5 minutes, 4 hours limit 200ug, multimodal analgesia: paracetamol 1000 mg iv every 6 hours until patient can take orally, change to 1000 mg orally every 6 hours total 3 days, Parecoxib 40 mg IV x 4 doses then COX2 inhibitor (etoricoxib 90 mg orally x2 days)
  Interventions: Procedure: Thoracic continuous epidural analgesia
- No CEA (Active Comparator): IV PCA fentanyl, IV patient-controlled analgesia; bolus mode only, fentanyl 15 ug/bolus, lockout interval 5 minutes, 4 hours limit 200ug multimodal analgesia: paracetamol 1000 mg IV every 6 hours until patient can take orally, change to 1000 mg orally q 6 hours total 3 days, Parecoxib 40 mg IV x 4 doses then COX2 inhibitor (Etoricoxib 90 mg orally x2 days)
  Interventions: Procedure: Thoracic continuous epidural analgesia

INTERVENTIONS:
Procedure: Thoracic continuous epidural analgesia — Continuous epidural catheter (Portex ™, Epidural Minipack , Smiths Medical), infused with 0.0625% bupivacaine (Marcaine™, Aspen Holdings) with morphine (morphine M&H™) 0.02 mg/ml 5 ml/h postoperative until POD3 morning Connected with The Sapphire ™ Infusion System Patient-Controlled-Analgesia (PCA) pump(fentanyl (fentanyl-Hameln™, Siam Bioscience): intravenous bolus mode only 15 ug/bolus, lockout interval 5 minutes, 4-hour limit 200 ug)
  Postoprative analgesia: intravenous paracetamol (infulgan ™, Yuria-Pharm), tablet paracetamol (SaRa ™), Parecoxib (Dynastat ™, Pfizer), Etoricoxib (Arcoxia ™, MSD)

SUMMARY:
This prospective randomized controlled study is aimed to determine the advantages of thoracic epidural analgesia for open upper abdominal surgery in combination with multimodal analgesia compared with no thoracic epidural analgesia on postoperative pain control. The primary outcome is total opioid consumption in postoperative 72 hours. Secondary outcomes are the success of continuous epidural analgesia or complications of this technique, pain intensity, morbidity and mortality compare to no continuous epidural analgesia.

DETAILED DESCRIPTION:
Continuous epidural analgesia (CEA) for open upper abdominal surgery has been showed the analgesic analgesia for open abdominal surgery. However the technical difficulty, complications especially hypotension, pruritus of CEA impede the popularity of technique compared to intravenous patient-controlled analgesia (IV PCA) in multimodal analgesia. This study is aimed to study of the role of CEA and multimodal analgesia in open abdominal surgery compare to IV PCA.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 years
* open upper abdominal surgery
* American Society of Anesthesiologists (ASA) grade I-III

Exclusion Criteria:

* contraindications to CEA
* inability communication
* patient's refusal
* emergency surgery
* BMI > 35

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
Amount of postoperative opioid consumption | postoperative 24 hours
  amount of fentanyl (microgram)
Amount of postoperative opioid consumption | postoperative 48 hours
  amount of fentanyl (microgram)
Amount of postoperative opioid consumption | postoperative 72 hours
  amount of fentanyl (microgram)

SECONDARY OUTCOMES:
Pain intensity | postoperative 6 hours until 72 hours postoperative
  numerical rating scale 0-10 (0= no pain, 10= worst pain)
Intraoperative opioid usage | intraoperative
  intravenous fentanyl consumption
Complications of thoracic epidural analgesia | postoperative 24 hours, 48 hours, 72 hours
  hypotension, pruritus
Percentage of patient to do out of bed activities | postoperative day 1
  standing beside the patient's bed
Length of hospital stay | days from patient admission until discharge, an average within 1 week
  hospital admission
Morbidity | Up to 30 days postoperative
  Myocardial ischemia, pneumonia, deep vein thrombosis
Mortality | Up to 30 days postoperative
  Death

CONTACTS AND LOCATIONS:
Overall Officials: Suwimon Tangwiwat, MD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Guay J, Nishimori M, Kopp SL. Epidural Local Anesthetics Versus Opioid-Based Analgesic Regimens for Postoperative Gastrointestinal Paralysis, Vomiting, and Pain After Abdominal Surgery: A Cochrane Review. Anesth Analg. 2016 Dec;123(6):1591-1602. doi: 10.1213/ANE.0000000000001628. PMID 27870743
- [Result] Salicath JH, Yeoh EC, Bennett MH. Epidural analgesia versus patient-controlled intravenous analgesia for pain following intra-abdominal surgery in adults. Cochrane Database Syst Rev. 2018 Aug 30;8(8):CD010434. doi: 10.1002/14651858.CD010434.pub2. PMID 30161292
- [Result] Greco KJ, Brovman EY, Nguyen LL, Urman RD. The Impact of Epidural Analgesia on Perioperative Morbidity or Mortality after Open Abdominal Aortic Aneurysm Repair. Ann Vasc Surg. 2020 Jul;66:44-53. doi: 10.1016/j.avsg.2019.10.054. Epub 2019 Oct 28. PMID 31672606
- [Result] Simpson RE, Fennerty ML, Colgate CL, Kilbane EM, Ceppa EP, House MG, Zyromski NJ, Nakeeb A, Schmidt CM. Post-Pancreaticoduodenectomy Outcomes and Epidural Analgesia: A 5-year Single-Institution Experience. J Am Coll Surg. 2019 Apr;228(4):453-462. doi: 10.1016/j.jamcollsurg.2018.12.038. Epub 2019 Jan 21. PMID 30677524
- [Result] Groen JV, Khawar AAJ, Bauer PA, Bonsing BA, Martini CH, Mungroop TH, Vahrmeijer AL, Vuijk J, Dahan A, Mieog JSD. Meta-analysis of epidural analgesia in patients undergoing pancreatoduodenectomy. BJS Open. 2019 Apr 29;3(5):559-571. doi: 10.1002/bjs5.50171. eCollection 2019 Oct. PMID 31592509